CLINICAL TRIAL: NCT01013792
Title: A Multi-centered, Prospective, Randomized, Double-blinded, Comparison of an Investigational Non-adherent Dressing to 3M Tegaderm Matrix Dressing With PHI Technology in the Management of Non-healing Diabetic Foot Ulcers
Brief Title: A Comparison of an Investigational Dressing to Tegaderm Matrix Wound Dressing in the Management of Diabetic Foot Ulcers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Expired study materials; low subject recruitment
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 05-011091
Record Dates: First submitted 2009-11-13; First posted 2009-11-16 (Estimated); Results first posted 2015-03-23 (Estimated); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Foot Ulcer, Diabetic
Keywords: Diabetic; Foot; Ulcer; Neuropathic; Tegaderm Matrix Dressing; DFU; Wound Care; PHI
MeSH Terms: conditions — Diabetic Foot; Ulcer | interventions — Bandages

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-adherent Wound Dressing (Experimental): The non-adherent dressing is the same as the Tegaderm Matrix dressing, with potassium chloride, rubidium chloride, calcium chloride, zinc chloride, potassium citrate and citric acid removed. This dressing is a Class I medical device (21 CFR Sec. 878.4020 Occlusive wound dressing) that is exempt from premarket notification procedures.
  Interventions: Device: Wound Dressing
- Tegaderm Matrix Dressing with PHI (Active Comparator): A commercial wound dressing to be used per manufacturer's instructions for use.
  Interventions: Device: Wound Dressing

INTERVENTIONS:
Device: Wound Dressing — Acetate mesh carrier with ointment (water, PEGs)
  Arms: Non-adherent Wound Dressing
Device: Wound Dressing — Acetate mesh carrier with ointment (water, PEGs, cations, citric acid)
  Arms: Tegaderm Matrix Dressing with PHI

SUMMARY:
The primary objective is to:

* Assess the effect of the Non-adherent study dressing to 3M Tegaderm Matrix Dressing with PHI technology on wound healing in patients with a diabetic foot ulcer.

Secondary objectives are to:

* Assess the adverse events that occur in subjects randomized to the investigational dressing in comparison to subjects randomized to the Tegaderm Matrix Dressing with PHI technology.
* Assess the costs of using the investigational dressing compared to the Tegaderm Matrix Dressing with PHI technology.
* Assess and compare the impact that these dressings have on patients' quality of life.
* Assess the wound's biological response and pH to the study dressings.

DETAILED DESCRIPTION:
The primary objective of this study is to compare the effect of an investigational, non-adherent dressing to a commercial wound dressing, 3M™ Tegaderm™ Matrix Dressing with PHI™ technology (Matrix dressing), in the management of diabetic foot ulcers. Subjects' wounds will be observed for a four week, pre-treatment period with wound assessments being made and samples of wound fluid and tissue collected and analyzed to characterize the wound. Following this pre-treatment observational stage, subjects continuing to meet inclusion/exclusion criteria will be randomly assigned, with stratification by center, wound size and wound duration, in either of two groups in the eight week treatment stage of the study. Subjects in one group will have their wound managed with an investigational non-adherent dressing, and subjects in the other group will have their wound managed with a Matrix dressing. At Visit 4 (start of the treatment stage of the study), subjects with a study wound that is less than 1 cm2 at this point will be dropped from the study. A second investigational device will be used to measure the pH of the wound, which will be compared to wound healing data.

Pre-treatment Stage Secondary Objectives

1. To measure and compare changes in wound size and wound assessments with changes in wound biomarker levels, wound pH, microbial load, and changes in systemic levels of C-reactive protein and homocysteine.
2. To measure and compare changes in wound biomarker levels, pH, and microbial load, and changes in systemic (blood) levels of C-reactive protein and homocysteine, looking for relationships.

Treatment Stage Secondary Objectives

1. To measure and compare the incidence of adverse events experienced by subjects in each of the 2 treatment groups.
2. To measure and compare the wound characteristics of each treatment group.
3. To measure and compare the subjects' quality of life of each treatment group.
4. To measure and compare the cost effectiveness of each treatment group.
5. To measure and compare changes in wound size with changes in wound biomarker levels, pH, and microbial load; and changes in systemic (blood) levels of C-reactive protein and homocysteine.
6. To measure and compare changes in wound biomarker levels, pH, microbial load, and changes in systemic levels of C-reactive protein and homocysteine, looking for relationships within treatment groups and overall.
7. To assess the ease of using these dressing

Post-treatment Stage Secondary Objectives

Subjects whose wounds heal prior to Visit 12 are expected to have a follow-up appointment 12-14 weeks after their wound has healed. Subjects whose wounds do not heal by Visit 12 are expected to complete a follow-up appointment 12-14 weeks after their last appointment. The objectives of this are to determine the frequency of complete healing between the two treatment groups and to determine the number of wounds that had healed by the end of the treatment phase and remained healed for each group at the follow-up appointment.

The objective is to measure and compare the percentage of wounds healed by Visit 12 (or before) that remained healed at the follow-up appointment by treatment group.

ELIGIBILITY:
Inclusion Criteria:

1. Is the subject 18 years of age or older?
2. Does the subject have a chronic full thickness diabetic foot ulcer (DFU) inferior to the malleolus that has been present for a minimum of four (4) weeks?
3. Does the diabetic foot ulcer measure greater than 1.0 cm2 and less than 25.0 cm2 after the wound is debrided?
4. Does the subject show evidence of neuropathy?
5. Is the subject's wound free of tunneling and showing no exposed periosteum or bone and free of clinical infection defined as the presence of local signs and symptoms including purulence, warmth, tenderness, pain, induration, cellulitis, bullae, crepitus, abscess, fasciitis and osteomyelitis?
6. Is the study wound able to be off loaded or achieve pressure relief and permit daily dressing changes?
7. Is the subject willing to have three (3) wound biopsies taken (Visit 0, 4 and 8)?
8. Is the subject willing to have photos taken of their wound and permit use of the photos in publications?
9. Has the subject or their legally authorized representative signed an Institutional Review Board approved informed consent document and authorized the use and disclosure of protected health information?
10. Does the subject have adequate circulation to the foot as evidenced by an Ankle Brachial Index (ABI) of 0.8 - 1.2; or if the ABI is greater than 1.2, does the subject show toe pressures >40 mmHg, or transcutaneous oximetry (TcPO2) > 40 mm Hg, or does the subject show adequate circulation on an arterial Doppler study? (ABI or Doppler results must be < 45 days old.)
11. Is the subject able to comply with the protocol requirements?
12. If the subject is a woman of child bearing potential is she practicing an acceptable form of birth control as determined by the Investigator, and is she willing to have a pregnancy test?

Exclusion Criteria:

1. Is the subject pregnant or breast feeding or have they given birth within the 3 weeks preceding the screening visit?
2. Has the subject been diagnosed with a malignant disease and received chemotherapy or treatment for a malignancy within the past 1 year?
3. Does the subject have an infection requiring systemic antibiotic treatment?
4. Has the subject ever received radiation therapy or other local therapy for malignancy at the extremity where the wound is located (from patient history)?
5. Is the subject currently using systemic steroids, or have they used systemic steroids within the previous 2 weeks, or are they projected to require systemic steroid use during the study as evidenced by a history of chronic systemic steroid use? (Topical steroids (except on the study extremity) and steroid inhalants will be allowed in the study.)
6. Does the subject have Lupus or Crohn's disease?
7. Does the subject have an oxygen dependency?
8. Has the subject received hyperbaric oxygen therapy within the previous 90 days?
9. Has the subject had vascular surgery relating to the wound within 30 days prior to the Screening Visit?
10. Does the subject have an active Charcot foot deformity of the foot presenting the ulcer?
11. Has the subject received Dermagraft®, Apligraf, or any other biologically active wound care product, or used Regranex Gel®, KGF, TGFβ or another topical growth factor to the study ulcer within the 30 days prior to the Screening visit?
12. Does the subject's wound require the use of topical silver, topical antibiotics, enzymatic debridement agents or other topical agents?
13. Has the subject been enrolled in any investigational study within 30 days of the Screening Visit?
14. Does the subject have any medical condition that in the opinion of the investigator should exclude him/her from participating in the study?
15. Has the subject received ultrasonic debridement or electrical stimulation within 7 days of the Screening Visit?

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph V Boykin, MD, Principal Investigator — HCA Retreat Hospital
Locations (6):
- United States (6):
  - Terry Treadwell, MD, Montgomery, Alabama
  - Alex Reyzelman, DPM, Castro Valley, California
  - Wyatt Payne, MD, Bay Pines, Florida
  - Vickie Driver, DPM, Boston, Massachusetts
  - William Marston, MD, Chapel Hill, North Carolina
  - Joseph Boykin, MD, Richmond, Virginia

REFERENCES:
- [Background] Schultz G, Mozingo D, Romanelli M, Claxton K. Wound healing and TIME; new concepts and scientific applications. Wound Repair Regen. 2005 Jul-Aug;13(4 Suppl):S1-11. doi: 10.1111/j.1067-1927.2005.1304S1.x. No abstract available. PMID 16008735
- [Background] Keast DH, Bowering CK, Evans AW, Mackean GL, Burrows C, D'Souza L. MEASURE: A proposed assessment framework for developing best practice recommendations for wound assessment. Wound Repair Regen. 2004 May-Jun;12(3 Suppl):S1-17. doi: 10.1111/j.1067-1927.2004.0123S1.x. PMID 15230830
- [Background] Mustoe T. Understanding chronic wounds: a unifying hypothesis on their pathogenesis and implications for therapy. Am J Surg. 2004 May;187(5A):65S-70S. doi: 10.1016/S0002-9610(03)00306-4. PMID 15147994
- [Background] Falanga V. The chronic wound: impaired healing and solutions in the context of wound bed preparation. Blood Cells Mol Dis. 2004 Jan-Feb;32(1):88-94. doi: 10.1016/j.bcmd.2003.09.020. PMID 14757419
- [Background] Xu L, McLennan SV, Lo L, Natfaji A, Bolton T, Liu Y, Twigg SM, Yue DK. Bacterial load predicts healing rate in neuropathic diabetic foot ulcers. Diabetes Care. 2007 Feb;30(2):378-80. doi: 10.2337/dc06-1383. No abstract available. PMID 17259515
- [Background] Blakytny R, Jude E. The molecular biology of chronic wounds and delayed healing in diabetes. Diabet Med. 2006 Jun;23(6):594-608. doi: 10.1111/j.1464-5491.2006.01773.x. PMID 16759300
- [Background] Steed DL. Wound-healing trajectories. Surg Clin North Am. 2003 Jun;83(3):547-55, vi-vii. doi: 10.1016/S0039-6109(02)00208-6. PMID 12822725
- [Background] Robson MC, Hill DP, Woodske ME, Steed DL. Wound healing trajectories as predictors of effectiveness of therapeutic agents. Arch Surg. 2000 Jul;135(7):773-7. doi: 10.1001/archsurg.135.7.773. PMID 10896369
- [Background] Margolis DJ, Gelfand JM, Hoffstad O, Berlin JA. Surrogate end points for the treatment of diabetic neuropathic foot ulcers. Diabetes Care. 2003 Jun;26(6):1696-700. doi: 10.2337/diacare.26.6.1696. PMID 12766096
- [Background] Gelfand JM, Hoffstad O, Margolis DJ. Surrogate endpoints for the treatment of venous leg ulcers. J Invest Dermatol. 2002 Dec;119(6):1420-5. doi: 10.1046/j.1523-1747.2002.19629.x. PMID 12485449
- [Background] Sheehan P, Jones P, Giurini JM, Caselli A, Veves A. Percent change in wound area of diabetic foot ulcers over a 4-week period is a robust predictor of complete healing in a 12-week prospective trial. Plast Reconstr Surg. 2006 Jun;117(7 Suppl):239S-244S. doi: 10.1097/01.prs.0000222891.74489.33. PMID 16799391
- [Background] Steed DL, Hill DP, Woodske ME, Payne WG, Robson MC. Wound-healing trajectories as outcome measures of venous stasis ulcer treatment. Int Wound J. 2006 Mar;3(1):40-7. doi: 10.1111/j.1742-4801.2006.00178.x. PMID 16650209
- [Background] Kantor J, Margolis DJ. A multicentre study of percentage change in venous leg ulcer area as a prognostic index of healing at 24 weeks. Br J Dermatol. 2000 May;142(5):960-4. doi: 10.1046/j.1365-2133.2000.03478.x. PMID 10809855
- [Background] Greener B, Hughes AA, Bannister NP, Douglass J. Proteases and pH in chronic wounds. J Wound Care. 2005 Feb;14(2):59-61. doi: 10.12968/jowc.2005.14.2.26739. No abstract available. PMID 15739652
- [Background] Karim RB, Brito BL, Dutrieux RP, Lassance FP, Hage JJ. MMP-2 assessment as an indicator of wound healing: A feasibility study. Adv Skin Wound Care. 2006 Jul-Aug;19(6):324-7. doi: 10.1097/00129334-200607000-00011. PMID 16885646
- [Background] Pirayesh A, Dessy LA, Rogge FJ, Hoeksema HJ, Sinove YM, Dall' Antonia A, Jawad MA, Gilbert PM, Rubino C, Scuderi N, Blondeel R, Monstrey S. The efficacy of a polyhydrated ionogen impregnated dressing in the treatment of recalcitrant diabetic foot ulcers: a multi-centre pilot study. Acta Chir Belg. 2007 Nov-Dec;107(6):675-81. doi: 10.1080/00015458.2007.11680145. PMID 18274183
- [Background] van Rossum M, Vooijs DP, Walboomers XF, Hoekstra MJ, Spauwen PH, Jansen JA. The influence of a PHI-5-loaded silicone membrane, on cutaneous wound healing in vivo. J Mater Sci Mater Med. 2007 Jul;18(7):1449-56. doi: 10.1007/s10856-006-0112-z. Epub 2007 Mar 27. PMID 17387598
- [Background] Schmidtchen A, Wolff H, Hansson C. Differential proteinase expression by Pseudomonas aeruginosa derived from chronic leg ulcers. Acta Derm Venereol. 2001 Nov-Dec;81(6):406-9. doi: 10.1080/000155501317208336. PMID 11859942
- [Background] Edwards JV, Howley PS. Human neutrophil elastase and collagenase sequestration with phosphorylated cotton wound dressings. J Biomed Mater Res A. 2007 Nov;83(2):446-54. doi: 10.1002/jbm.a.31171. PMID 17477392
- [Background] Rushton I. Understanding the role of proteases and pH in wound healing. Nurs Stand. 2007 Apr 18-24;21(32):68, 70, 72 passim. doi: 10.7748/ns2007.04.21.32.68.c4499. PMID 17479791
- [Background] Gethin GT, Cowman S, Conroy RM. The impact of Manuka honey dressings on the surface pH of chronic wounds. Int Wound J. 2008 Jun;5(2):185-94. doi: 10.1111/j.1742-481X.2007.00424.x. PMID 18494624 (Retraction: PMID 24827812 Int Wound J. 2014 Jun;11(3):342)
- [Background] Wysocki AB, Staiano-Coico L, Grinnell F. Wound fluid from chronic leg ulcers contains elevated levels of metalloproteinases MMP-2 and MMP-9. J Invest Dermatol. 1993 Jul;101(1):64-8. doi: 10.1111/1523-1747.ep12359590. PMID 8392530
- [Background] Ravanti L, Kahari VM. Matrix metalloproteinases in wound repair (review). Int J Mol Med. 2000 Oct;6(4):391-407. PMID 10998429
- [Background] Muller M, Trocme C, Lardy B, Morel F, Halimi S, Benhamou PY. Matrix metalloproteinases and diabetic foot ulcers: the ratio of MMP-1 to TIMP-1 is a predictor of wound healing. Diabet Med. 2008 Apr;25(4):419-26. doi: 10.1111/j.1464-5491.2008.02414.x. PMID 18387077
- [Background] Schonfelder U, Abel M, Wiegand C, Klemm D, Elsner P, Hipler UC. Influence of selected wound dressings on PMN elastase in chronic wound fluid and their antioxidative potential in vitro. Biomaterials. 2005 Nov;26(33):6664-73. doi: 10.1016/j.biomaterials.2005.04.030. PMID 15978664
- [Background] Veves A, Sheehan P, Pham HT. A randomized, controlled trial of Promogran (a collagen/oxidized regenerated cellulose dressing) vs standard treatment in the management of diabetic foot ulcers. Arch Surg. 2002 Jul;137(7):822-7. doi: 10.1001/archsurg.137.7.822. PMID 12093340
- [Background] Smeets R, Ulrich D, Unglaub F, Woltje M, Pallua N. Effect of oxidised regenerated cellulose/collagen matrix on proteases in wound exudate of patients with chronic venous ulceration. Int Wound J. 2008 Jun;5(2):195-203. doi: 10.1111/j.1742-481X.2007.00367.x. PMID 18494625
- [Background] Lobmann R, Zemlin C, Motzkau M, Reschke K, Lehnert H. Expression of matrix metalloproteinases and growth factors in diabetic foot wounds treated with a protease absorbent dressing. J Diabetes Complications. 2006 Sep-Oct;20(5):329-35. doi: 10.1016/j.jdiacomp.2005.08.007. PMID 16949521
- [Background] Fasciglione GF, Marini S, D'Alessio S, Politi V, Coletta M. pH- and temperature-dependence of functional modulation in metalloproteinases. A comparison between neutrophil collagenase and gelatinases A and B. Biophys J. 2000 Oct;79(4):2138-49. doi: 10.1016/S0006-3495(00)76461-7. PMID 11023917
- [Background] Nwomeh BC, Liang HX, Cohen IK, Yager DR. MMP-8 is the predominant collagenase in healing wounds and nonhealing ulcers. J Surg Res. 1999 Feb;81(2):189-95. doi: 10.1006/jsre.1998.5495. PMID 9927539

RESULTS

PARTICIPANT FLOW:
Groups:
- Tegaderm Matrix Dressing With PHI Technology: Wound Dressing: Acetate mesh carrier with ointment (water, PEGs, cations, citric acid)
Period: Overall Study
Arm/Group | Non-adherent Wound Dressing | Tegaderm Matrix Dressing With PHI Technology
Started | 14 | 16
Completed | 12 | 11
Not Completed | 2 | 5
Not completed — Study suspended | 2 | 1
Not completed — Adverse Event | 0 | 3
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: All subjects had diabetic foot ulcers between 1.0cm2 and 25.0cm2 at randomization
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-adherent Wound Dressing | Tegaderm Matrix Dressing With PHI Technology | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (7.06) | 54.1 (11.01) | 56.9 (9.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 12 | 12 | 24
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 0 | 1
  Black or African American | 1 | 3 | 4
  Hispanic or Latino | 0 | 3 | 3
  White | 12 | 10 | 22
Region of Enrollment [Number; unit: participants]
  United States | 14 | 16 | 30
Diabetic foot ulcer area [Median (Full Range); unit: cm2] | 3.1 [1.3 to 11.3] | 2.8 [1.1 to 14.6] | 2.8 [1.1 to 14.6]
Diabetic foot ulcer age [Number; unit: participants]
  4-12 weeks | 3 | 3 | 6
  13-26 weeks | 4 | 2 | 6
  27-52 weeks | 1 | 1 | 2
  >1-5 years | 4 | 10 | 14
  >5 years | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent Diabetic Foot Ulcer Area Reduction From Baseline to Last Treatment Visit
Description: A positive value indicates a reduction in area relative to baseline, while a negative value indicates an increase in area relative to baseline (at time of randomization), calculated as [(Baseline - Week 8)/Baseline] x 100%.
Time Frame: up to 8 weeks
Population: All participants that are randomized
Measure: Median (Full Range); unit: percent change of baseline area
Arm/Group | Non-adherent Wound Dressing | Tegaderm Matrix Dressing With PHI Technology
Number analyzed (Participants) | 14 | 16
percent change of baseline area | 18.1 [-70 to 100] | 34.2 [-43.9 to 100]

ADVERSE EVENTS:
Time Frame: 25 Weeks
Description: Start at patient consent/screening, through 4-week run-in, through 8 weeks treatment, through 12 weeks post-treatment follow-up
Arm/Group | Non-adherent Wound Dressing | Tegaderm Matrix Dressing With PHI Technology
Serious Adverse Events (participants affected / at risk) | 1/14 | 3/16
Other Adverse Events (participants affected / at risk) | 6/14 | 11/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-adherent Wound Dressing (N=14) | Tegaderm Matrix Dressing With PHI Technology (N=16)
Ischemic event with associate foot infection (Vascular disorders) | 0 (0) | 1 (1)
Ulcer/foot infection (Infections and infestations) | 1 (1) | 2 (2)
Subendocardial myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) — Renal failure, resulting in hemodialysis
Death (General disorders) | 1 (1) | 0 (0) — Unexpected death in his sleep
Bladder Cancer (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-adherent Wound Dressing (N=14) | Tegaderm Matrix Dressing With PHI Technology (N=16)
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) — Upper respiratory infection
Wound/Skin Infection (Infections and infestations) | 4 (8) | 7 (9) — Infection/Cellulitis in wound or periwound skin
Pain, Trauma, Blister (Skin and subcutaneous tissue disorders) | 5 (7) | 6 (8)
Phlebitis, Edema, Swelling (Vascular disorders) | 2 (2) | 2 (3)
Abdominal Pain (Gastrointestinal disorders) | 2 (3) | 1 (1)
Bleeding (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypoglycemia (Endocrine disorders) | 0 (0) | 1 (2) — Dizzy spells
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Surgical resection (Surgical and medical procedures) | 1 (1) | 1 (1)
Sprained ankle (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other